CLINICAL TRIAL: NCT02389374
Title: A Study to Assess Safety of Current Standard Malaria Treatment and an Assessment of Glucose-6-dehydrogenase Status in South-east Bangladesh
Brief Title: A Study to Assess Safety of Current Standard Malaria Treatment and an Assessment of G6PD Status in South-east Bangladesh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-14053
Record Dates: First submitted 2015-02-05; First posted 2015-03-17 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Chloroquine; Artemether, Lumefantrine Drug Combination; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- chloroquine primaquine 14days (Other): P.vivax malaria patients receiving chloroquine and primaquine 14days as per guidelines
  Interventions: Drug: chloroquine; Drug: Primaquine
- artemether-lumefantrine primaquine 1day (Other): P.falciparum malaria patients receiving artemether-lumefantrine combination and primaquine 1day as per guidelines
  Interventions: Drug: Artemether-lumefantrine combination; Drug: Primaquine
- artemether-lumefantrine primaquine 14days (Other): mixed malaria infection receiving artemether-lumefantrine combination and primaquine 14days as per guidelines
  Interventions: Drug: Artemether-lumefantrine combination; Drug: Primaquine

INTERVENTIONS:
Drug: chloroquine — standard dose
  Arms: chloroquine primaquine 14days
Drug: Artemether-lumefantrine combination — standard dose
  Arms: artemether-lumefantrine primaquine 14days; artemether-lumefantrine primaquine 1day
Drug: Primaquine — single dose
  Arms: artemether-lumefantrine primaquine 1day
Drug: Primaquine — 14 days
  Arms: artemether-lumefantrine primaquine 14days; chloroquine primaquine 14days

SUMMARY:
This is a study assessing safety and efficacy of current national guidelines for the treatment of uncomplicated malaria in Bangladesh as well as to assess the G6PD status among the enrolled patients.

DETAILED DESCRIPTION:
The national guidelines for the treatment of uncomplicated malaria in Bangladesh currently recommend a standard dose of artemether-lumefantrine followed by a single dose of primaquine for P. falciparum malaria and a three day course of chloroquine followed by 14 days of primaquine for vivax malaria.Currently the national treatment guidelines do not include any testing for G6PD deficiency before treatment with primaquine. In order to guarantee safe and efficacious treatment for all patients diagnosed with uncomplicated malaria in Bangladesh, it is essential to monitor the effectiveness and safety of the recommended treatment guidelines. This trial therefore evaluates the local efficacy and safety of the current first line treatment and assesses the G6PD status of the enrolled patients.

Patients with uncomplicated malaria attending the health care center, who meet the study inclusion criteria will be enrolled, treated on site and followed up for 28 days. The follow-up will consist of a fixed schedule of check-up visits and corresponding clinical and laboratory examinations. The study will provide efficacy data for both artemether-lumefantrine and chloroquine and will generate data on G6PD status in the region, which will provide vital information for policy makers in regards to the wider roll out of primaquine for the radical cure of vivax malaria.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 months
* P. vivax or P. falciparum monoinfection or P.v. / P.f. mixed infection
* Presence of axillary temperature ≥ 37.5°C or history of fever during the past 24 hrs
* Ability to swallow oral medication.
* Ability and willingness to comply with the study protocol for the duration of the study
* Informed consent/assent from the patient or from a parent or guardian in the case of children.

Exclusion Criteria:

* Presence of general danger signs in children aged under 5 years or signs of severe malaria according to the definitions of WHO
* Presence of severe malnutrition
* Acute anaemia <8g/dL
* Regular medication, which may interfere with antimalarial pharmacokinetics
* History of hypersensitivity reactions or contraindications to any of the drug(s) tested or used as alternative treatment(s)
* A positive pregnancy test or lactating

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

REFERENCES:
- [Derived] Alam MS, Ley B, Nima MK, Johora FT, Hossain ME, Thriemer K, Auburn S, Marfurt J, Price RN, Khan WA. Molecular analysis demonstrates high prevalence of chloroquine resistance but no evidence of artemisinin resistance in Plasmodium falciparum in the Chittagong Hill Tracts of Bangladesh. Malar J. 2017 Aug 15;16(1):335. doi: 10.1186/s12936-017-1995-5. PMID 28806961
- [Derived] Ley B, Alam MS, Thriemer K, Hossain MS, Kibria MG, Auburn S, Poirot E, Price RN, Khan WA. G6PD Deficiency and Antimalarial Efficacy for Uncomplicated Malaria in Bangladesh: A Prospective Observational Study. PLoS One. 2016 Apr 29;11(4):e0154015. doi: 10.1371/journal.pone.0154015. eCollection 2016. PMID 27128675

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Started | 55 | 115 | 11
Completed | 46 | 87 | 10
Not Completed | 9 | 28 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days | Total
Number analyzed (Participants) | 55 | 115 | 11 | 181
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 18 [11 to 27] | 22 [14 to 30] | 14 [7 to 26] | 20 [11 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 6 | 46
  Male | 36 | 94 | 5 | 135
Region of Enrollment [Number; unit: participants]
  Bangladesh | 55 | 115 | 11 | 181

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Adverse and Serious Adverse Events Following Unsupervised Primaquine Treatment
Description: The proportion of adverse and serious adverse events following unsupervised primaquine treatment until day 28
Time Frame: during follow up (day 28)
Measure: Number; unit: events
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Number analyzed (Participants) | 55 | 115 | 11
events | 0 | 0 | 0

2. Secondary Outcome: Proportion of Patients Receiving Blood Transfusion and With Severe Anaemia (Hb<7g/dl)
Time Frame: day 28
Measure: Number; unit: participants
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Number analyzed (Participants) | 55 | 115 | 11
participants | 0 | 0 | 0

3. Secondary Outcome: Fractional Change in Hb Between Baseline and Day 9 and 16
Time Frame: day 0 and 16
Measure: Mean (95% Confidence Interval); unit: percent change Hb
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Number analyzed (Participants) | 55 | 115 | 11
percent change Hb
  baseline to day 9 | -2.3 [-6.2 to 1.5] | -7.7 [-11.2 to -4.2] | -13.8 [-22.1 to -5.5]
  baseline to day 16 | -0.5 [-6.1 to 5.1] | NA [NA to NA] — No visit on day 16 | -8.3 [-20.2 to 3.7]

4. Secondary Outcome: Proportion of Patients With Anaemia Less Than 8g/dl on Day 2
Time Frame: on day 2
Measure: Number; unit: participants with Hb under 8g/dl
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Number analyzed (Participants) | 55 | 115 | 11
participants with Hb under 8g/dl | 0 | 2 | 0

5. Secondary Outcome: Proportion of Patients With Any Parasitemia on Day 3 After Treatment
Time Frame: day 3
Measure: Number; unit: participants
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Number analyzed (Participants) | 55 | 115 | 11
participants | 0 | 2 | 0

6. Secondary Outcome: Proportion of Patients With Fever on Day 2 After Treatment
Time Frame: day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Number analyzed (Participants) | 55 | 112 | 11
Participants | 0 | 0 | 0

7. Secondary Outcome: Recurrence of Parasitaemia Within 16 Days of Follow up
Time Frame: day 16
Measure: Number; unit: Recurrences of Parsitaemia
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Number analyzed (Participants) | 55 | 115 | 11
Recurrences of Parsitaemia | 0 | 0 | 0

8. Secondary Outcome: Proportion of Patients Adhering to 14 Days of Primaquine Treatment in the Vivax Cohort as Measured by Pill Count
Time Frame: day 16
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Number analyzed (Participants) | 43 | 115 | 9
Participants | 34 | NA — this outcome was only collected for the other two arms | 7

9. Secondary Outcome: The Distribution of G6PD Activity Measured in U/gHb Among All Malaria Patients
Time Frame: day 0
Measure: Median (Inter-Quartile Range); unit: U/gHb
Groups:
- All Malaria Patients: single Arm/Group for all participants
Arm/Group | All Malaria Patients
Number analyzed (Participants) | 181
U/gHb | 7.82 [6.62 to 10.00]

10. Secondary Outcome: Frequency and Type of Variants of the G6PD Gene Within the Study Population
Description: Frequency and type of variants of the G6PD gene within the study population
Time Frame: day 0 or 1
Population: data were not collected
Arm/Group | All Malaria Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Chloroquine Primaquine 14days | Artemether-lumefantrine Primaquine 1day | Artemether-lumefantrine Primaquine 14days
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/115 | 0/11
Other Adverse Events (participants affected / at risk) | 0/55 | 0/115 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No